CLINICAL TRIAL: NCT04048746
Title: Evaluation of the Written Information Delivered by the General Practitioner of the Patients Presenting to the Emergency Room for an Aggravation of Asthma
Acronym: ASTHMAVILLE
Status: Terminated | Type: Observational
Why Stopped: The PI decided to stop.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ASTHMAVILLE
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ASTHMA: The patient presents to the emergency department for an aggravation of his asthma. The patient later sees an emergency investigator for medical care for his aggravation of asthma. When the patient's condition is stabilized, the investigator checks his eligibility for study and offers to participate. If the patient agrees, the investigator gives him the questionnaire and possibly helps to fill it out.
  When the investigator returns to see the patient for a reassessment of his condition, he retrieves the completed questionnaire. He verifies that the patient has completed the questionnaire. Prescriptions and action plans are retrieved by the principal investigator either in digitized format from the patient's computerized medical record or in paper format. Each medication prescription and each action plan are read by the principal investigator and evaluated according to the grids.

SUMMARY:
Asthma is a common pathology (prevalence 6.4% in 2018, in France), currently managed by the general practitioner in general practice. It is a chronic disease at risk of exacerbation, which can lead to the use of care. The treatment of asthma is based on a basic treatment, to be taken every day, the purpose of which is to avoid acute exacerbations and lead a normal life. There is also an emergency treatment, to be taken in case of sudden worsening of the respiratory state. The asthmatic patient is the first actor in his care. He must be able to react in case of emergency. A good knowledge of the disease and its treatment as well as training in self-management of crises are thus fundamental and must be part of its medical care. The existence of an exacerbation represents a criterion of non-control of the disease, thus a failure of the long-term care of the patient. The optimization of this care includes individual issues aimed at improving the quality of life and collective by reducing the avoidable use of care and thus the expenses related to this disease. It relies on therapeutic education sessions as well as the provision of written information, clear and detailed by the doctor. This information consists of the writing of a detailed medication prescription as well as the dispensing of a written action plan.

The action plan must describe the actions to be taken by the patient in case of exacerbation of his asthma, to regain control. Regarding the format, it can be coupled to the prescription drug (action plan and prescription on the same prescription) or distinct from the prescription drug (a prescription for drugs and a prescription for the action plan). In some countries, "ready-to-use" action plans have been validated by learned societies, which is not the case today in France. In Canada, a study demonstrated in 2006 that 46% of asthmatic patients followed in hospital had an action plan, while the national average was estimated at about 10% in 2010. There is little data in France on the proportion of patients with asthma action plans.

Unlike the action plan, which is little distributed to the patient, the prescription drug for asthma is always given to the patient at the end of the consultation and specifies the procedures for taking treatments.

As part of this work, the investigators are interested in evaluating the written information given to the adult asthmatic patient by their general practitioner: the action plan but also the prescription medication.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Asthma patient
* Emergency Patient Counselor for GHPSJ for management of worsening asthma
* Patient followed for his asthma in town by a general practitioner
* Francophone patient

Exclusion Criteria:

* Patient opposing his participation in the study
* Patient under tutorship or curatorship
* Patient deprived of liberty
* Patient under safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthma patient consulting the Emergencies of the GHPSJ for the management of a worsening of his asthma
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Written action plan | Day 1
  This oucome measure the percentage of included patients who have received a written action plan from their general practitioner who follows them for their asthma regardless of the format (separate or part of the same prescription as the prescription drug).

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Salmeron, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France